CLINICAL TRIAL: NCT03255642
Title: Efficacy and Safety of Melatonin and Rivotril Treatment for Idiopathic Rapid Eye Movement Sleep Disorder: Prospective Randomized Study.
Brief Title: Efficacy and Safety of Melatonin and Clonazepam for IRBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Won Chul Shin, Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-03-011
Record Dates: First submitted 2017-05-29; First posted 2017-08-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Clonazepam; Melatonin; Treatment; REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — Melatonin; Clonazepam

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open-label study
Who Masked: Outcomes Assessor
Masking Description: Mask treatment arm when analyzing polysomnography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin 2mg (Active Comparator): 4 weeks of 2mg of prolonged release Melatonin
  Interventions: Drug: Melatonin 2mg
- ClonazePAM 0.5 MG (Placebo Comparator): 4 weeks of 0.5mg of rivotril
  Interventions: Drug: ClonazePAM 0.5 MG

INTERVENTIONS:
Drug: Melatonin 2mg — 4 weeks of 2mg prolonged release melatonin (Circadin)
  Other Names: Circadin
  Arms: Melatonin 2mg
Drug: ClonazePAM 0.5 MG — 4 weeks of 0.5mg clonazepam (Rivotril)
  Other Names: Rivotril
  Arms: ClonazePAM 0.5 MG

SUMMARY:
This study aimed to evaluate influence of melatonin or clonazepam treatment on symptom and polysomnographic parameters in patients with idiopathic REM sleep behavior disorder.

DETAILED DESCRIPTION:
This study is open-label parallel trial with 4 weeks treatment with slow-release melatonin (Circadin) or with clonazepam (Rivotril).

Polysomnography, symptom diary and questionnaire (Clinical Global Impression, RBDQ-HK, PSQI, ESS, SSS, ISI, BDI-II) will be performed before and after 4 weeks of each medications.

ELIGIBILITY:
Inclusion Criteria:

* REM sleep behavior disorder (ICSD-3 criteria)

Exclusion Criteria:

* Neurological disorder including epilepsy or stroke
* History of psychiatric illness
* Neurodegenerative disease including dementia or parkinsonism.
* Medication affecting sleep within 1 month
* Intake of melatonin or clonazepam within 1 week.
* Unable to complete questionnaires

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Automated REM without atonia index | 4 weeks of prolonged release melatonin 2mg or clonazepam 0.5mg
  Percentage seconds with chin EMG amplitude<1uV/ Total REM seconds.

SECONDARY OUTCOMES:
Clinical Global Impression of RBD symptom severity | 4 weeks of prolonged release melatonin 2mg or clonazepam 0.5mg
  Clinical Global Impression scale score provided by patient and caregiver.
REM sleep behavior disorder symptom severity | 4 weeks of prolonged release melatonin 2mg or clonazepam 0.5mg
  REM sleep behavior disorder questionnaire-Hong Kong total score
Sleep quality | 4 weeks of prolonged release melatonin 2mg or clonazepam 0.5mg
  Pittsburg Sleep Quality Index total score
Depression | 4 weeks of prolonged release melatonin 2mg or clonazepam 0.5mg
  Beck depression inventory-II total score

CONTACTS AND LOCATIONS:
Overall Officials: Won Chul Shin, M.D. Ph.D., Principal Investigator — KyungHee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferri R, Marelli S, Ferini-Strambi L, Oldani A, Colli F, Schenck CH, Zucconi M. An observational clinical and video-polysomnographic study of the effects of clonazepam in REM sleep behavior disorder. Sleep Med. 2013 Jan;14(1):24-9. doi: 10.1016/j.sleep.2012.09.009. Epub 2012 Oct 23. PMID 23098778
- [Background] Kunz D, Mahlberg R. A two-part, double-blind, placebo-controlled trial of exogenous melatonin in REM sleep behaviour disorder. J Sleep Res. 2010 Dec;19(4):591-6. doi: 10.1111/j.1365-2869.2010.00848.x. PMID 20561180
- [Background] McCarter SJ, Boswell CL, St Louis EK, Dueffert LG, Slocumb N, Boeve BF, Silber MH, Olson EJ, Tippmann-Peikert M. Treatment outcomes in REM sleep behavior disorder. Sleep Med. 2013 Mar;14(3):237-42. doi: 10.1016/j.sleep.2012.09.018. Epub 2013 Jan 23. PMID 23352028
- [Background] McGrane IR, Leung JG, St Louis EK, Boeve BF. Melatonin therapy for REM sleep behavior disorder: a critical review of evidence. Sleep Med. 2015 Jan;16(1):19-26. doi: 10.1016/j.sleep.2014.09.011. Epub 2014 Oct 13. PMID 25454845
- [Background] Nardone R, Golaszewski S, Holler Y, Christova M, Trinka E, Brigo F. Neurophysiological insights into the pathophysiology of REM sleep behavior disorders: a review. Neurosci Res. 2013 Jul;76(3):106-12. doi: 10.1016/j.neures.2013.03.009. Epub 2013 Mar 28. PMID 23542221
- [Background] Iranzo A, Molinuevo JL, Santamaria J, Serradell M, Marti MJ, Valldeoriola F, Tolosa E. Rapid-eye-movement sleep behaviour disorder as an early marker for a neurodegenerative disorder: a descriptive study. Lancet Neurol. 2006 Jul;5(7):572-7. doi: 10.1016/S1474-4422(06)70476-8. PMID 16781987
- [Derived] Byun JI, Shin YY, Seong YA, Yoon SM, Hwang KJ, Jung YJ, Cha KS, Jung KY, Shin WC. Comparative efficacy of prolonged-release melatonin versus clonazepam for isolated rapid eye movement sleep behavior disorder. Sleep Breath. 2023 Mar;27(1):309-318. doi: 10.1007/s11325-022-02572-8. Epub 2022 Feb 9. PMID 35141811